CLINICAL TRIAL: NCT05242757
Title: Clinical Study on the Safety and Efficacy of Mixed-activated Killer Immune Cells in the Treatment of Primary Hepatocellular Carcinoma
Brief Title: Clinical Study of MAK Immune Cells in the Treatment of PHC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Zhongnan Hospital
Record Dates: First submitted 2021-12-14; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-11

CONDITIONS: Primary Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To evaluate the safety and reliminary efficacy of MAK immune cells in the treatment of PHC. (Experimental): To evaluate the safety and reliminary efficacy of MAK immune cells in the treatment of primary hepatocellular carcinoma.
  Interventions: Other: Mixed-activated Killer Immune Cells

INTERVENTIONS:
Other: Mixed-activated Killer Immune Cells — Mixed-activated Killer Immune Cells Peripheral intravenous infusion therapy

SUMMARY:
The investigators will plan to recruit 20 patients with liver cancer CNLC stage Ⅲa and Ⅲb who are older than 18 years old. Peripheral blood mononuclear cells were obtained and then the MAK(Mixed-activated Killer) cells were injected, and then the safety and efficacy were observed.

DETAILED DESCRIPTION:
The investigators will plan to recruit 20 patients with liver cancer CNLC stage Ⅲa and Ⅲb who are older than 18 years old. Peripheral venous blood was collected twice (50-60ml/time, 2 times, 1 week apart) from each patient. Peripheral blood mononuclear cells were separated, induced, expanded, and cultured in vitro for a total of 1 week to obtain physiological conditions Immune cell populations with tumor-killing activity (mainly MAK immune cells mainly CD3-CD16 + CD56 + and CD3 + CD56 +), and then the MAK(Mixed-activated Killer) cells were injected intravenously for three days. Observe that the patient received cell therapy 24h, The safety and efficacy of 1 month, 2 months, and 3 months, and monitoring of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old, regardless of gender.
2. Patients with primary hepatocellular carcinoma.
3. According to the "Regulations for Diagnosis and Treatment of Primary Liver Cancer (2019 Edition)" by the Health Commission of the People's Republic of China Liver cancer staging scheme, patients with Ⅲa and Ⅲb.
4. The expected survival time is ≥6 months.
5. Peripheral blood white blood cell count ≥3×10^9 /L.
6. Understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Patients with immunodeficiency or autoimmune diseases (such as rheumatoid arthritis, systemic lupus erythematosus, multiple Primary sclerosis, insulin dependent diabetes, etc.).
2. Patients with a history of other malignant tumors in the past 5 years.
3. Patients who participated in other clinical trials or clinical research treatments within 3 months before this clinical study By.
4. Patients who have received other cell therapy within the past 6 months.
5. Patients with fever who have not effectively controlled the infection.
6. Patients with high allergies or a history of severe allergies.
7. Patients who are allergic to albumin.
8. Patients after organ transplantation; patients who have been using or are using immunosuppressive agents for a long time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Detecting the dynamic changes of circulating tumor cell count ( > 4 CTC counts per milliliter of blood acted as positive ) | three months
  Peripheral blood was collected 6 times at baseline, 24 hours after two MAK cell transfusions, and 1, 2, and 3 months after the last MAK cell transfusions to detect the changes in the number of circulating tumor cells ( > 4 CTC counts per milliliter of blood acted as positive ).
The size (tumor diameter) and number (tumor recurrence lesions) of PHC tumors were examined by enhanced abdominal CT | three months
  At baseline and 1, 2 and 3 months after the last cell transfusion, a total of 4 abdominal enhanced CT examinations were performed to count the tumor size (tumor diameter) and number of tumor recurrence lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Ye, MD, PHD, Study Chair — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Hubei, Wuhan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morotti M, Albukhari A, Alsaadi A, Artibani M, Brenton JD, Curbishley SM, Dong T, Dustin ML, Hu Z, McGranahan N, Miller ML, Santana-Gonzalez L, Seymour LW, Shi T, Van Loo P, Yau C, White H, Wietek N, Church DN, Wedge DC, Ahmed AA. Promises and challenges of adoptive T-cell therapies for solid tumours. Br J Cancer. 2021 May;124(11):1759-1776. doi: 10.1038/s41416-021-01353-6. Epub 2021 Mar 29. PMID 33782566